CLINICAL TRIAL: NCT02018315
Title: Clinical Trial of Citric Acid Cycle Stimulation in Energy-deficiency States: Treatment Development for Glucose Transporter Type I Deficiency Syndrome (G1D) (NMTUT 2010B)
Brief Title: Treatment Development for Glucose Transporter Type I Deficiency Syndrome (G1D)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juan Pascual (Other)
Responsible Party: Sponsor-Investigator, Juan Pascual, Associate Professor, Director of the Rare Brain Disorders Program, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UTSW 122010-186
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome; GLUT1 Deficiency Syndrome
Keywords: G1D; Glut1 Disorder; Glucose Transporter Type 1 Disorder; Glucose Transporter Type I Disorder
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triheptanoin (Experimental): Triheptanoin (C7 oil, liquid) dosed at 1 g/kg body weight divided and administered 4 times per day via mouth or g-tube for 3 months.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin is a 7-carbon medium chain triglyceride
  Other Names: C7; Heptanoate

SUMMARY:
The purpose of this trial is to determine if an alternative energy source will impact brain metabolism in a disorder characterized by glucose metabolism failure in the brain.

The central hypothesis tested in this investigation is whether circumventing impaired glucose metabolism is feasible, safe and potentially promising by supplying anaplerotic precursors through metabolism of odd-carbon fatty acids that can enter the citric acid cycle (CAC) through alternative metabolic pathways.

DETAILED DESCRIPTION:
Triheptanoin, a nutritional supplement long used in other metabolic disorders and also added to foods and cosmetics, will be used to complement any diet that G1D patients may be receiving at enrollment with the exception of the ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 1 month to <21 years of age
* Diagnosed with glucose transporter type I deficiency.
* Age matched (within 1 year) controls not diagnosed with G1D.

Exclusion Criteria:

* All subjects carrying body metal implants incompatible with the exposure to a magnetic field
* Subjects unable to tolerate the MRI and MRS procedures due to anxiety
* Subjects receiving oxygen supplementation or those confined to a bed or stretcher
* Subjects currently receiving a ketogenic diet, due to a high risk of seizure recurrence while transitioning off ketosis.
* Patients behaviorally unable to hold still for imaging procedures (rather than limited by seizure activity) will be excluded.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. Pascual, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Marin-Valencia I, Good LB, Ma Q, Duarte J, Bottiglieri T, Sinton CM, Heilig CW, Pascual JM. Glut1 deficiency (G1D): epilepsy and metabolic dysfunction in a mouse model of the most common human phenotype. Neurobiol Dis. 2012 Oct;48(1):92-101. doi: 10.1016/j.nbd.2012.04.011. Epub 2012 Apr 23. PMID 22683290
- [Background] Marin-Valencia I, Roe CR, Pascual JM. Pyruvate carboxylase deficiency: mechanisms, mimics and anaplerosis. Mol Genet Metab. 2010 Sep;101(1):9-17. doi: 10.1016/j.ymgme.2010.05.004. Epub 2010 Jun 9. PMID 20598931
- [Background] Wang D, Sands T, Tang M, Monani U, De Vivo D. Glucose Transporter Type 1 Deficiency Syndrome. 2002 Jul 30 [updated 2025 Mar 6]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1430/ PMID 20301603
- [Background] Perez-Duenas B, Prior C, Ma Q, Fernandez-Alvarez E, Setoain X, Artuch R, Pascual JM. Childhood chorea with cerebral hypotrophy: a treatable GLUT1 energy failure syndrome. Arch Neurol. 2009 Nov;66(11):1410-4. doi: 10.1001/archneurol.2009.236. PMID 19901175
- [Background] Pascual JM, Campistol J, Gil-Nagel A. Epilepsy in inherited metabolic disorders. Neurologist. 2008 Nov;14(6 Suppl 1):S2-S14. doi: 10.1097/01.nrl.0000340787.30542.41. PMID 19225367
- [Background] Pascual JM, Wang D, Hinton V, Engelstad K, Saxena CM, Van Heertum RL, De Vivo DC. Brain glucose supply and the syndrome of infantile neuroglycopenia. Arch Neurol. 2007 Apr;64(4):507-13. doi: 10.1001/archneur.64.4.noc60165. Epub 2007 Feb 12. PMID 17296829
- [Background] Pascual JM, Wang D, Lecumberri B, Yang H, Mao X, Yang R, De Vivo DC. GLUT1 deficiency and other glucose transporter diseases. Eur J Endocrinol. 2004 May;150(5):627-33. doi: 10.1530/eje.0.1500627. PMID 15132717
- [Background] Pascual JM, Wang D, Yang R, Shi L, Yang H, De Vivo DC. Structural signatures and membrane helix 4 in GLUT1: inferences from human blood-brain glucose transport mutants. J Biol Chem. 2008 Jun 13;283(24):16732-42. doi: 10.1074/jbc.M801403200. Epub 2008 Apr 3. PMID 18387950
- [Background] Pascual JM. [Glucose transport hereditary diseases]. Med Clin (Barc). 2006 Nov 11;127(18):709-14. doi: 10.1157/13095099. Spanish. PMID 17169300
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Mao X, Cheng J, Yoo J, Noebels JL, De Vivo DC. A mouse model for Glut-1 haploinsufficiency. Hum Mol Genet. 2006 Apr 1;15(7):1169-79. doi: 10.1093/hmg/ddl032. Epub 2006 Feb 23. PMID 16497725
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Jhung S, Sun RP, De Vivo DC. Glut-1 deficiency syndrome: clinical, genetic, and therapeutic aspects. Ann Neurol. 2005 Jan;57(1):111-8. doi: 10.1002/ana.20331. PMID 15622525
- [Background] Pascual JM, Lecumberri B, Wang D, Yang R, Engelstad K, De Vivo DC. [Type 1 glucose transporter (Glut1) deficiency: manifestations of a hereditary neurological syndrome]. Rev Neurol. 2004 May 1-15;38(9):860-4. Spanish. PMID 15152356
- [Background] Wang D, Pascual JM, Iserovich P, Yang H, Ma L, Kuang K, Zuniga FA, Sun RP, Swaroop KM, Fischbarg J, De Vivo DC. Functional studies of threonine 310 mutations in Glut1: T310I is pathogenic, causing Glut1 deficiency. J Biol Chem. 2003 Dec 5;278(49):49015-21. doi: 10.1074/jbc.M308765200. Epub 2003 Sep 16. PMID 13129919
- [Background] Pascual JM, Van Heertum RL, Wang D, Engelstad K, De Vivo DC. Imaging the metabolic footprint of Glut1 deficiency on the brain. Ann Neurol. 2002 Oct;52(4):458-64. doi: 10.1002/ana.10311. PMID 12325075
- [Background] Iserovich P, Wang D, Ma L, Yang H, Zuniga FA, Pascual JM, Kuang K, De Vivo DC, Fischbarg J. Changes in glucose transport and water permeability resulting from the T310I pathogenic mutation in Glut1 are consistent with two transport channels per monomer. J Biol Chem. 2002 Aug 23;277(34):30991-7. doi: 10.1074/jbc.M202763200. Epub 2002 May 24. PMID 12032147
- [Background] De Vivo DC, Wang D, Pascual JM, Ho YY. Glucose transporter protein syndromes. Int Rev Neurobiol. 2002;51:259-88. doi: 10.1016/s0074-7742(02)51008-4. No abstract available. PMID 12420362
- [Background] Brockmann K, Wang D, Korenke CG, von Moers A, Ho YY, Pascual JM, Kuang K, Yang H, Ma L, Kranz-Eble P, Fischbarg J, Hanefeld F, De Vivo DC. Autosomal dominant glut-1 deficiency syndrome and familial epilepsy. Ann Neurol. 2001 Oct;50(4):476-85. doi: 10.1002/ana.1222. PMID 11603379

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Triheptanoin: Triheptanoin (C7 oil, liquid) dosed at 1 g/kg body weight divided and administered 4 times per day via mouth or g-tube for 3 months.
Period: Overall Study
Arm/Group | Experimental: Triheptanoin
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Triheptanoin
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] — Confirm that 2 subjects were enrolled that were older than 20 years of age. Inclusion criteria was not updated to reflect this change in enrollment.
  Years | 12.5 [2 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in Spike-wave Fraction of the EEG Recording Time
Description: Visual analysis of EEG recording to determine the fraction of spike-range within the area of recording.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Triheptanoin
Number analyzed (Participants) | 14
Participants | 13

2. Secondary Outcome: Number of Participants With Change in Brain Metabolic Rate After 3 Months
Description: Magnetic Resonance Imaging (MRI) used to calculate brain metabolic rate. Brain metabolic rate compared before oil ingestion (Baseline), 90 minutes after oil ingestion, and after 3 months of daily oil ingestion in each participant. Triheptanoin metabolism may lead to increased oxygen consumption only while the brain undergoes a reduction of ictogenesis. We hypothesize that when ictogenesis is abolished by triheptanoin or absent at baseline, triheptanoin exerts little or no effect on CMR02.
Time Frame: 3 months
Population: 5 participants out of the 14 total participants enrolled completed the optional MRI . Reasons for participants electing to not participate in imaging included inability to remain immobile due to movement disorder or anxiety, immaturity, metal implants, and personal choice.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Triheptanoin
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Arm/Group | Triheptanoin
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triheptanoin (N=14)
Gastric discomfort (Gastrointestinal disorders) | 1
weight gain (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes